CLINICAL TRIAL: NCT00403234
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Pilot Study to Evaluate the Analgesic Efficacy of BTDS on Postoperative Pain During Rehabilitation Following Total Knee Arthroplasty
Brief Title: Safety of Buprenorphine Transdermal System (BTDS) in Subjects With Acute Postoperative Pain After Total Knee Replacement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to administrative reasons not related to efficacy or safety.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP2003
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; opioid; transdermal; TKA (total knee arthroplasty)
MeSH Terms: conditions — Pain, Postoperative | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BTDS 10 (Experimental): Buprenorphine transdermal patch 10 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal patch
- BTDS 20 (Experimental): Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal patch
- BTDS 30 (Experimental): Buprenorphine transdermal patch 30 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal patch
- Placebo TDS (Placebo Comparator): Placebo patches were similar to BTDS 10 and 20.
  Interventions: Drug: Placebo BTDS

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 10 mcg/h applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS 10
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS 20
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patches 10 mcg/h and 20 mcg/h (total of 30 mcg/h) applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS 30
Drug: Placebo BTDS — Placebo to match BTDS transdermal 10 and 20 patches applied for 7-day wear.
  Arms: Placebo TDS

SUMMARY:
The objectives in this study are to evaluate: (1) efficacy of buprenorphine transdermal system (BTDS, Butrans™) on postoperative pain following total knee replacement surgery; (2) the impact of BTDS on functional rehabilitative measures after total knee replacement surgery; and 3) the safety of BTDS after total knee replacement surgery. The double-blind treatment period is for 28 days during which time supplemental analgesic medication will be provided to all subjects in addition to study drug.

Purdue Pharma L.P. terminated the trial early due to administrative reasons not related to efficacy or safety. The focus of this study became safety evaluations.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 18 to 80 years of age with American Society of Anesthesiologists (ASA) physical status classification of 1, 2 or 3
* Scheduled to undergo unilateral total knee arthroplasty (TKA) for the treatment of the osteoarthritis.

Exclusion Criteria:

* Subjects who have pain or disability in a site other than the operative joint.
* Subjects who have had total knee arthroplasty within 6 months of the scheduled surgery or are scheduled to undergo bilateral knee arthroplasty.
* Subjects whose body mass index (BMI) is 40 or more.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Accurate Clinical Trials, Inc, San Clemente, California
  - Southeastern Clinical Research Consultants, Orlando, Florida
  - Greater Chesapeake Orthopaedic Associates, Baltimore, Maryland
  - Sewickley Valley Hospital, Sewickley, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: 02-Nov-2006 (first patient first visit) to 20-Apr-2007 (last patient last visit) at 5 medical/research centers in the US.
  The study was terminated early due to reasons unrelated to efficacy or safety.
Pre-assignment Details: Enrolled: N = 14. Following surgery and recovery from anesthesia, subjects had to demonstrate moderate to severe pain within 6 hours postsurgery ("Pain Right Now" rating of ≥ 2 on a 4-point scale where 0 = no pain and 3 = severe pain), then their intravenous patient-controlled analgesia morphine device was activated. N = 10 were randomized.
Groups:
- Placebo: Placebo transdermal patch applied for 7-day wear.
- BTDS 30: Buprenorphine transdermal patch 10 + 20 mcg/h applied for 7-day wear
Period: Overall Study
Arm/Group | Placebo | BTDS 10 | BTDS 20 | BTDS 30
Started | 2 | 3 | 3 | 2
Completed | 1 | 2 | 2 | 2
Not Completed | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BTDS 10 | BTDS 20 | BTDS 30 | Total
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (8.49) | 58.3 (7.37) | 66.3 (4.04) | 59 (7.07) | 62.6 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 2 | 8
  Male | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety
Description: Adverse Events that occurred after the signing of the informed consent up to end of study and 7 days after, discontinuation, or SAEs occurring up to 30 days following the last study visit were followed until the AE resolved.
Time Frame: From signed informed consent to 7 days after end of study (approx. 35 days)
Population: The Safety Population consisted of subjects who were randomized, received at least 1 dose of double-blind study drug and had at least 1 safety assessment during double-blind treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | BTDS 10 | BTDS 20 | BTDS 30
Number analyzed (Participants) | 2 | 3 | 3 | 2
participants
  Deaths | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Serious Adverse Events | 0 | 0 | 0 | 0
  All Other Adverse Events in ≥ 4.5% of subjects | 2 | 2 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are recorded up to 7 days after the last dose or until the last visit. Ongoing AEs at the last visit are followed until resolution or for 30 days after the visit. Serious AEs are followed until resolution or the event stabilize.
Description: AEs were learned of through spontaneous reports and subject interview.
Arm/Group | Placebo | BTDS 10 | BTDS 20 | BTDS 30
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3 | 3/3 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | BTDS 10 (N=3) | BTDS 20 (N=3) | BTDS 30 (N=2)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 1 — Systematic and nonsystematic assessment
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 — Systematic and nonsystematic assessment
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 — Systematic and nonsystematic assessment
Chest pain (General disorders) | 0 | 1 | 0 | 0 — Systematic and nonsystematic assessment
Chills (General disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Pyrexia (General disorders) | 0 | 1 | 0 | 2 — Systematic and nonsystematic assessment
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Systematic and nonsystematic assessment
Gamma-Glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 — Systematic and nonsystematic assessment
Oxygen saturation decreased (Investigations) | 0 | 0 | 2 | 0 — Systematic and nonsystematic assessment
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — Systematic and nonsystematic assessment
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Systematic and nonsystematic assessment
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Systematic and nonsystematic assessment
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 — Systematic and nonsystematic assessment
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 — Systematic and nonsystematic assessment
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Hallucinations (Psychiatric disorders) | 0 | 0 | 1 | 0 — Systematic and nonsystematic assessment
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 — Systematic and nonsystematic assessment
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Systematic and nonsystematic assessment
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Systematic and nonsystematic assessment

LIMITATIONS AND CAVEATS:
This trial was terminated early due to administrative reasons not related to efficacy or safety. The efficacy data are not presented since the objective of this study was changed prior to study unblinding, identifying it as a safety study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days